CLINICAL TRIAL: NCT02670473
Title: Clinical Performance of Existing Wearers of Enfilcon A Following a Refit With Fanfilcon A Lenses for 4 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-55 (CV-15-09)
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- enfilcon A (habitual) (No Intervention): Participants are habitual wearers of enfilcon A lens and refitted with fanfilcon A lens.
- fanfilcon A (test) (Experimental): Participants are habitual wearers of enfilcon A lens and refitted with fanfilcon A lens.
  Interventions: Device: fanfilcon A (test)

INTERVENTIONS:
Device: fanfilcon A (test) — contact lens
  Arms: fanfilcon A (test)

SUMMARY:
The aim of this dispensing study is to evaluate the clinical performance of habitual wearers of enfilcon A lenses following a refit with fanfilcon A lenses over 4 weeks of daily wear.

DETAILED DESCRIPTION:
This is a 30 subject, prospective, dispensing, bilateral wear, subject-masked study, reviewing the refit characteristics in a group of enfilcon A wearers switched to the fanfilcon A lens. Subject's habitual enfilcon A lenses will be evaluated at the first vist and then re-fitted with a pair of fanfilcon A lenses for 4 weeks of daily wear. After the dispensing visit, subjects will return for evaluations at 1 week, 2 weeks, and 4 weeks.

ELIGIBILITY:
Inclusion criteria

A person is eligible for inclusion in the study if he/she:

* Is between 18 and 40 years of age
* Has had a self-reported visual exam in the last two years
* Is an adapted enfilcon A contact lens wearer (at least 2 weeks in enfilcon A lens)
* Has a contact lens spherical prescription between -1.00 to - 6.00
* Has a spectacle cylinder up to 0.75D (Diopters) in each eye.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood, and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria

A person will be excluded from the study if he/she:

* Is not a habitual wearer of enfilcon A lenses
* Has a CL (Contact Lens) prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder ≥1.00D of cylinder in either eye.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 3-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montés-Mico, O.D., PhD, Principal Investigator — Optometry Research Group (GIO) University of Valencia
Locations (1):
- Optometry Research Group (GIO) Optics Department, University of Valencia, Valencia, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Participants: Participants are habitual wearers of enfilcon A lens and refitted with fanfilcon A lens.
  fanfilcon A (test): contact lens
Period: Overall Study
Arm/Group | Overall Participants
Started | 35
Completed | 34
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 34 subjects completed the study and included in the baseline analysis.
Arm/Group | Overall Participants
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.15 (5.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Lens Fit - Centration
Description: Lens fit evaluation of centration for enfilcon A habitual lens (control) is assessed at baseline and fanfilcon A lens (test) is assessed at 1 week, 2 weeks, and 4 weeks. Scale: optimum, decentration acceptable, decentration unacceptable.
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Measure: Number; unit: percentage of eyes
Groups:
- Habitual Lenses: Baseline: enfilcon A habitual lens (control)
- Fanfilcon A: 1 Week; Fanfilcon A: 2 Weeks; Fanfilcon A: 4 Weeks: fanfilcon A lens (test)
Arm/Group | Habitual Lenses: Baseline | Fanfilcon A: 1 Week | Fanfilcon A: 2 Weeks | Fanfilcon A: 4 Weeks
Number analyzed (Participants) | 35 | 35 | 34 | 34
percentage of eyes
  Optimum | 88 | 97 | 99 | 100
  Decentration acceptable | 12 | 3 | 1 | 0
  Decentration unacceptable | 0 | 0 | 0 | 0

2. Primary Outcome: Lens Fit - Post-blink Movement
Description: Lens fit evaluation of post-blink movement for enfilcon A habitual lens (control) is assessed at baseline and fanfilcon A lens (test) is assessed at 1 week, 2 weeks, and 4 weeks. Scale 0-5 Likert scale, 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement.
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Measure: Number; unit: percentage of eyes
Arm/Group | Habitual Lenses: Baseline | Fanfilcon A: 1 Week | Fanfilcon A: 2 Weeks | Fanfilcon A: 4 Weeks
Number analyzed (Participants) | 35 | 35 | 34 | 34
percentage of eyes
  Insufficient, unacceptable movement | 0 | 0 | 0 | 0
  Minimal, but acceptable movement | 1 | 1 | 0 | 0
  Optimal movement | 35 | 3 | 6 | 18
  Moderate, but acceptable movement | 64 | 96 | 91 | 79
  Excessive, unacceptable movement | 0 | 0 | 3 | 3

3. Primary Outcome: Lens Tightness on Push-up
Description: Lens fit evaluation of tightness on push-up test for enfilcon A habitual lens (control) is assessed at baseline and fanfilcon A lens (test) is assessed at 1 week, 2 weeks, and 4 weeks. Scale: 0%-100%, 0%=Falls from cornea without lid support, 50%=Optimum, 100%=No movement.
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of lens tightness
Arm/Group | Habitual Lenses: Baseline | Fanfilcon A: 1 Week | Fanfilcon A: 2 Weeks | Fanfilcon A: 4 Weeks
Number analyzed (Participants) | 35 | 35 | 34 | 34
percentage of lens tightness | 50 (5) | 49 (2) | 50 (3) | 50 (3)

4. Primary Outcome: Overall Fit Acceptance
Description: Overall fit acceptance for enfilcon A habitual lens (control) is assessed at baseline and fanfilcon A lens (test) is assessed at 1 week, 2 weeks, and 4 weeks. Scale 0-4, 0=Should not be worn, 1=Borderline but unacceptable, 2=Minimum acceptable, early review, 3=Not perfect but okay to dispense, 4=Perfect.
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Measure: Number; unit: percentage of eyes
Arm/Group | Habitual Lenses: Baseline | Fanfilcon A: 1 Week | Fanfilcon A: 2 Weeks | Fanfilcon A: 4 Weeks
Number analyzed (Participants) | 35 | 35 | 34 | 34
percentage of eyes
  Should not be worn | 0 | 0 | 0 | 0
  Borderline but unacceptable | 0 | 0 | 0 | 0
  Minimum acceptable | 0 | 0 | 0 | 0
  Not perfect but okay | 9 | 0 | 7 | 3
  Perfect | 91 | 100 | 93 | 97

5. Secondary Outcome: Overall Comfort
Description: Subjective rating of overall comfort for enfilcon A habitual lens (control) is assessed at baseline and fanfilcon A lens (test) is assessed at 1 week, 2 weeks, and 4 weeks. Scale 0-10, 0=could feel, 10=cannot feel.
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Habitual Lenses: Baseline | Fanfilcon A: 1 Week | Fanfilcon A: 2 Weeks | Fanfilcon A: 4 Weeks
Number analyzed (Participants) | 35 | 35 | 34 | 34
units on a scale | 8.03 (0.97) | 8.91 (1.06) | 8.97 (0.83) | 8.85 (0.96)

6. Secondary Outcome: Dryness Overall
Description: Subjective rating of overall dryness for enfilcon A habitual lens (control) is assessed at baseline and fanfilcon A lens (test) is assessed at 1 week, 2 weeks, and 4 weeks. Scale 0-10, 0=very dry, 10=no dryness.
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Habitual Lenses: Baseline | Fanfilcon A: 1 Week | Fanfilcon A: 2 Weeks | Fanfilcon A: 4 Weeks
Number analyzed (Participants) | 35 | 35 | 34 | 34
units on a scale | 7.88 (1.32) | 8.82 (1.09) | 8.85 (1.08) | 8.82 (0.94)

7. Secondary Outcome: Handling
Description: Subjective rating of handling for enfilcon A habitual lens (control) is assessed at baseline and fanfilcon A lens (test) is assessed at 1 week, 2 weeks, and 4 weeks. Scale 0-10, 0=very difficult to handle, 10=very easy to handle.
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Habitual Lenses: Baseline | Fanfilcon A: 1 Week | Fanfilcon A: 2 Weeks | Fanfilcon A: 4 Weeks
Number analyzed (Participants) | 35 | 35 | 34 | 34
units on a scale | 8.85 (1.37) | 9.26 (1.16) | 9.59 (0.78) | 9.62 (0.74)

8. Secondary Outcome: Overall Vision Satisfaction
Description: Subjective rating of overall vision satisfaction for enfilcon A habitual lens (control) is assessed at baseline and fanfilcon A lens (test) is assessed at 1 week, 2 weeks, and 4 weeks. Scale 0-10, 0=very dissatisfied, 10=very satisfied.
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Habitual Lenses: Baseline | Fanfilcon A: 1 Week | Fanfilcon A: 2 Weeks | Fanfilcon A: 4 Weeks
Number analyzed (Participants) | 35 | 35 | 34 | 34
units on a scale | 9.24 (0.82) | 9.56 (0.79) | 9.79 (0.41) | 9.74 (0.51)

9. Secondary Outcome: Overall Satisfaction
Description: Subjective rating of overall satisfaction for enfilcon A habitual lens (control) at baseline and fanfilcon A lens (test) at 1 week, 2 weeks, and 4 weeks. Scale 1-4, 1=completely satisfied, 2=somewhat satisfied, 3=somewhat dissatisfied, 4=completely dissatisfied.
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Population: One participant withdrew from the study after week 1.
Measure: Number; unit: percentage of subjects
Arm/Group | Completely Satisfied | Somewhat Satisfied | Somewhat Dissatisfied | Completely Dissatisfied
Number analyzed (Participants) | 35 | 35 | 35 | 35
percentage of subjects
  Baseline - enfilcon A habitual lens (control) | 26 | 71 | 3 | 0
  1 week - fanfilcon A lens (test) | 53 | 47 | 0 | 0
  2 weeks - fanfilcon A lens (test): number analyzed (Participants) | 34 | 34 | 34 | 34
  2 weeks - fanfilcon A lens (test) | 65 | 35 | 0 | 0
  4 weeks - fanfilcon A lens (test): number analyzed (Participants) | 34 | 34 | 34 | 34
  4 weeks - fanfilcon A lens (test) | 71 | 29 | 0 | 0

10. Secondary Outcome: Lens Preference Overall
Description: Subject's overall preference for one of two contact lenses. Forced choice: enfilcon A habitual lens (control) or fanfilcon A lens (test).
Time Frame: 1 week, 2 weeks, and 4 weeks
Population: One participant withdrew from the study after week 1.
Measure: Number; unit: percentage of subjects
Groups:
- Habitual Lenses: enfilcon A habitual lens (control)
- Fanfilcon A Lens (Test): fanfilcon A lens (test)
Arm/Group | Habitual Lenses | Fanfilcon A Lens (Test)
Number analyzed (Participants) | 35 | 35
percentage of subjects
  1 week | 18 | 82
  2 weeks: number analyzed (Participants) | 34 | 34
  2 weeks | 6 | 94
  4 weeks: number analyzed (Participants) | 34 | 34
  4 weeks | 6 | 94

11. Secondary Outcome: Wearing Times
Description: Average wearing time and comfortable wearing times for enfilcon A habitual lens (control) is assessed at baseline and fanfilcon A lens (test) is assessed at 1 week, 2 weeks, and 4 weeks measured by hours.
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Habitual Lenses: Baseline | Fanfilcon A: 1 Week | Fanfilcon A: 2 Weeks | Fanfilcon A: 4 Weeks
Number analyzed (Participants) | 35 | 35 | 34 | 34
hours
  Average wearing time | 8.79 (1.67) | 9.82 (2.11) | 9.65 (1.69) | 9.85 (1.56)
  Comfortable wearing time | 7.65 (1.50) | 8.97 (2.44) | 8.91 (1.73) | 8.97 (1.40)

12. Secondary Outcome: Conjunctival Staining
Description: Conjunctival staining for enfilcon A habitual lens (control) is assessed at baseline and fanfilcon A lens (test) is assessed at 1 week, 2 weeks, and 4 weeks. (Scale 0-4, 0.5 steps 0=normal, 4=severe).
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Measure: Number; unit: percentage of eyes
Arm/Group | Habitual Lenses: Baseline | Fanfilcon A: 1 Week | Fanfilcon A: 2 Weeks | Fanfilcon A: 4 Weeks
Number analyzed (Participants) | 35 | 35 | 34 | 34
percentage of eyes
  0 | 100 | 97 | 99 | 94
  0.5 | 0 | 3 | 1 | 6
  1.0 | 0 | 0 | 0 | 0
  1.5 | 0 | 0 | 0 | 0
  2.0 | 0 | 0 | 0 | 0
  2.5 | 0 | 0 | 0 | 0
  3.0 | 0 | 0 | 0 | 0
  3.5 | 0 | 0 | 0 | 0
  4.0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Corneal Staining
Description: Corneal staining for enfilcon A habitual lens (control) is assessed at baseline and fanfilcon A lens (test) is assessed at 1 week, 2 weeks, and 4 weeks. Scale 0-4, 0.5 steps 0=normal, 4=severe.
Time Frame: Baseline, 1 week, 2 weeks, and 4 weeks
Measure: Number; unit: percentage of eyes
Arm/Group | Habitual Lenses: Baseline | Fanfilcon A: 1 Week | Fanfilcon A: 2 Weeks | Fanfilcon A: 4 Weeks
Number analyzed (Participants) | 35 | 35 | 34 | 34
percentage of eyes
  0 | 100 | 100 | 100 | 100
  0.5 | 0 | 0 | 0 | 0
  1.0 | 0 | 0 | 0 | 0
  1.5 | 0 | 0 | 0 | 0
  2.0 | 0 | 0 | 0 | 0
  2.5 | 0 | 0 | 0 | 0
  3.0 | 0 | 0 | 0 | 0
  3.5 | 0 | 0 | 0 | 0
  4.0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Overall Participants
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other